CLINICAL TRIAL: NCT05600101
Title: Development of Avatar-based Intervention to Support Patients Undergoing Reduced-Intensity Allogenic Stem Cell Transplantation
Brief Title: Development and Piloting an Avatar-based Intervention to Support Patients Undergoing Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Gregory A. Abel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-412; R44CA236253 (NIH)
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Hematopoietic Cell Transplantation
Keywords: Reduced intensity conditioning allogeneic transplant; Stem cell transplantation; Avatar-based technology; Artificial intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- care.coach Pilot (Experimental): The research study procedures include screening for eligibility, a brief call with a research assistant after tablet is given to subject, and a survey after a subject has completed the study.
  * 3 consecutive cohorts of 6 RIC HCT patients each.
  * care.coach is a "human-in the-loop" conversational agent (avatar) used to interact and converse with patients through natural dialogue and text-to-speech software that is powered by a team of trained human staff, called health advocates. A subject uses the avatar for up to 3 weeks.
  Interventions: Behavioral: Care.Coach

INTERVENTIONS:
Behavioral: Care.Coach — Care.coach is a "human-in the-loop" conversational agent (avatar) used to interact and converse with patients through natural dialogue and text-to-speech software that is powered by a team of trained human staff, called health advocates.

SUMMARY:
The goal of this research study is to provide an avatar-based technology during a subject's stay for participants who have been admitted to the hospital for reduced-intensity conditioning (RIC) allogeneic transplant. The intervention received will be the care.coach technology.

DETAILED DESCRIPTION:
This research study is a Pilot Study, which means the investigators are studying the application in a smaller group of people to understand whether the technology, care.coach, is easy to use.

This is a single site study at Dana-Farber Brigham and Women's Cancer Center.

* Aim 1 of the study will be an 8 - 10 participant focus group of nurses, navigator nurses, physicians, and NPs/PAs to refine the avatar protocols.
* Aim 2 of the study will be a pilot of 18 participants undergoing RIC allogeneic HCT in the hospital.

  * The research study procedures include screening for eligibility, a brief call with a research assistant during use of care.coach avatar, and a survey after study completion.
  * The avatar is designed to communicate with participants regarding transplantation education and provide reminders for eating, drinking, and activity.
  * care.coach is a digital, avatar-based technology that communicates using natural speech software.
  * care.coach is supporting this research by providing Dana-Farber access to its technology. The National Cancer Institute (NCI) also supports this research.

ELIGIBILITY:
Inclusion Criteria for HCT focus group:

* Age 18+.
* DFCI/HCC HCT nurse navigators, inpatient HCT nurses, and HCT physicians and extenders (NP/PA).

Inclusion Criteria for care.coach pilot:

* Age 18+.
* Admitted for reduced-intensity conditioning (RIC) allogeneic HCT

Exclusion Criteria for care.coach pilot:

Deemed by clinical staff or RA to be unable to converse with an avatar, due to:

* Severe, uncorrectable hearing impairment and simultaneous severe, uncorrectable vision impairment.
* Severe speech impairment that precludes understanding by staff (and by extension, by the avatar).
* Not fluent in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Abel, MPH, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted by a trained research assistant (RA) utilizing HIPAA-compliant and DFCI IRB approved patient approach procedures.
  A total of 18 participants were consented. Patients were approached and consented upon inpatient admission for RIC HCT. Patients were consented beginning on 12/6/2022 through 5/3/2023.
Pre-assignment Details: There were no significant events in the study for any patients between their enrollment and assignment to an arm or group of the study.
Groups:
- Care.Coach Pilot: The research study procedures include screening for eligibility, a brief call with a research assistant after tablet is given to subject, and a survey after a subject has completed the study.
  * 3 consecutive cohorts of 6 RIC HCT patients each.
  * care.coach is a "human-in the-loop" conversational agent (avatar) used to interact and converse with patients through natural dialogue and text-to-speech software that is powered by a team of trained human staff, called health advocates. A subject uses the avatar for up to 3 weeks.
  Care.Coach: Care.coach is a "human-in the-loop" conversational agent (avatar) used to interact and converse with patients through natural dialogue and text-to-speech software that is powered by a team of trained human staff, called health advocates.
- AI HCT Focus Group: A structured focus group arm consisted of HCT nurse navigators, inpatient HCT nurses, and HCT physicians. Participants provided their perspectives on patient facing artificial intelligence technology which was used to inform care.coach software protocols. Participation was limited to a single 60 minute focus group. The group consisted of of 2 bedside registered nurses, 1 oncology nurse, 3 transplant physicians, 1 physical therapist, 1 transplant nurse practitioner, 1 physician assistant transplant educator, and 1 nurse transplant educator.
Period: Overall Study
Arm/Group | Care.Coach Pilot | AI HCT Focus Group
Started | 18 | 10
Completed | 18 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: care.coach Pilot arm participants were patients admitted for inpatient RIC HCT. AI HCT Focus Group arm participants were HCT clinicians. Demographics cannot be reported for the AI HCT Focus Group arm participants as it was an anonymous focus group. No post-baseline Primary and Secondary Outcome Measure data were collected the AI HCT Focus Group.
Groups:
- AI HCT Focus Group: A structured focus group arm consisted of HCT nurse navigators, inpatient HCT nurses, and HCT physicians. Participants provided their perspectives on patient facing artificial intelligence technology which was used to inform care.coach software protocols. Participation was limited to a single 60 minute focus group.
- Total: Total of all reporting groups
Arm/Group | Care.Coach Pilot | AI HCT Focus Group | Total
Number analyzed (Participants) | 18 | 10 | 28
Age, Categorical [Count of Participants; unit: Participants] — Population: AI HCT Focus Group participant demographics were not analyzed.
  Participants
    number analyzed (Participants) | 18 | 0 | 18
    <=18 years | 0 |  | 0
    Between 18 and 65 years | 11 |  | 11
    >=65 years | 7 |  | 7
Sex: Female, Male [Count of Participants; unit: Participants] — Population: AI HCT Focus Group Participants demographics were not analyzed.
  Participants
    number analyzed (Participants) | 18 | 0 | 18
    Female | 11 |  | 11
    Male | 7 |  | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: AI HCT Focus Group participants demographics were not analyzed
  Participants
    number analyzed (Participants) | 18 | 0 | 18
    American Indian or Alaska Native | 0 |  | 0
    Asian | 2 |  | 2
    Native Hawaiian or Other Pacific Islander | 0 |  | 0
    Black or African American | 1 |  | 1
    White | 13 |  | 13
    More than one race | 0 |  | 0
    Unknown or Not Reported | 2 |  | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Retained
Description: Participants complete study protocol, including post-completion survey, from enrollment to hospital discharge or 3 weeks from enrollment (whichever is earlier).
Time Frame: Baseline to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Care.Coach Pilot
Number analyzed (Participants) | 18
Participants | 18

2. Secondary Outcome: Final Cohort Dissatisfaction Rate
Description: Percent of patients dissatisfied with the avatar in the third 6-patient cohort.
Time Frame: 3 weeks
Measure: Number; unit: percentage of particpants
Groups:
- Third Patient Cohort: Consisting of 6 participants, this cohort consisted of patients undergoing RIC HCT in the inpatient setting, consented as per the study protocol.
Arm/Group | Third Patient Cohort
Number analyzed (Participants) | 6
percentage of particpants | 0

3. Secondary Outcome: The Completion Rate Post-Pilot Survey
Description: Rate of completion of post-pilot survey within 1 week of discharge
Time Frame: 3 weeks
Measure: Number; unit: Survey Completion Rate Percentage
Arm/Group | Care.Coach Pilot
Number analyzed (Participants) | 18
Survey Completion Rate Percentage | 72

ADVERSE EVENTS:
Time Frame: For the care.coach Pilot arm participants, their adverse event data was collected from enrollment to hospital discharge or 3 weeks from enrollment (whichever was earlier). Adverse Events were not monitored or assessed for AI HCT Focus Group arm participants because there was no intervention.
Description: The definitions of adverse event and/or serious adverse event, used to collect adverse event information, did not differ from the clinicaltrials.gov definitions for the care.coach Pilot arm. Adverse Event data were not collected for the AI HCT Focus Group arm.
Groups:
- Focus Group Participants: A structured focus group arm consisted of HCT nurse navigators, inpatient HCT nurses, and HCT physicians. Participants provided their perspectives on patient facing artificial intelligence technology which was used to inform care.coach software protocols. Participation was limited to a single 60 minute focus group.
Arm/Group | Care.Coach Pilot | Focus Group Participants
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/0
Other Adverse Events (participants affected / at risk) | 0/18 | 0/0

LIMITATIONS AND CAVEATS:
This is a small cohort so results may need to be confirmed in a larger cohort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT05600101/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT05600101/ICF_001.pdf